CLINICAL TRIAL: NCT06062069
Title: A Phase 2, Double-Blind, Randomized, Placebo-Controlled Study to Evaluate the Efficacy, Safety, Tolerability, and Pharmacokinetics of CT-868 Administered for 16 Weeks to Overweight and Obese Adult Participants With Type 1 Diabetes Mellitus
Brief Title: A Study of CT-868 in Type 1 Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Carmot Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CT-868-004
Record Dates: First submitted 2023-09-14; First posted 2023-10-02 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Overweight; Obese; Type 1 Diabetes Mellitus
MeSH Terms: conditions — Overweight; Obesity; Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- CT-868 Low Dose (Experimental): Participants in this arm will receive the drug CT-868 in a subcutaneous injection form. The dosage is set at up to 1.8 mg, and it will be administered once daily for a total duration of 16 weeks.
  Interventions: Drug: CT-868; Device: CT-868 Pen Injector
- CT-868 Medium Dose (Experimental): Participants in this arm will receive the drug CT-868 in a subcutaneous injection form. The dosage is set at up to 4.1 mg, and it will be administered once daily for a total duration of 16 weeks.
  Interventions: Drug: CT-868; Device: CT-868 Pen Injector
- CT-868 High Dose (Experimental): Participants in this arm will receive the drug CT-868 in a subcutaneous injection form. The dosage is set at up to 6.6 mg, and it will be administered once daily for a total duration of 16 weeks.
  Interventions: Drug: CT-868; Device: CT-868 Pen Injector
- CT-868 Placebo (Placebo Comparator): Participants in this arm will receive a placebo designed to match the appearance and formulation of the drug CT-868. The intervention consists of a subcutaneous injection of this placebo. The placebo will be administered once daily for a duration of 16 weeks.
  Interventions: Device: CT-868 Pen Injector; Drug: CT-868 Pen Injector, Placebo

INTERVENTIONS:
Drug: CT-868 — CT-868 is an investigational medication administered subcutaneously via a pre-filled pen injector device.
  Arms: CT-868 High Dose; CT-868 Low Dose; CT-868 Medium Dose
Device: CT-868 Pen Injector — The CT-868 pen injector is a multi-dose, single-participant, disposable pen.
Drug: CT-868 Pen Injector, Placebo — The placebo pen injector is identical and contains the same ingredients except for CT-868.
  Arms: CT-868 Placebo

SUMMARY:
This study will evaluate the changes in glycemic control in overweight and obese adults with Type 1 Diabetes Mellitus after receiving CT-868 for 16 weeks. The effectiveness and safety of CT-868 will be compared to placebo. All participants will continue with their standard diabetes care using either an insulin pump (CSII) or multiple daily injections (MDI). Alongside their designated treatment, participants will receive guidance on managing their diabetes, including monitoring blood glucose levels and diet and exercise recommendations. Treatment assignments, either CT-868 plus insulin or placebo plus insulin will be randomly determined.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 years of age or older at the time of signing informed consent
* Have a documented clinical diagnosis of T1DM greater than or equal to 1 year before the Screening Visit
* Body mass index greater than or equal to27.0 kg/m2
* Hemoglobin A1c (HbA1c) level between 7.0% and 10.0%, inclusive, at the Screening Visit

Exclusion Criteria:

* Diagnosis of Type 2 diabetes mellitus (T2DM) or any other types of diabetes, except T1DM
* Experienced diabetic ketoacidosis (DKA) within 3 months prior to the Screening Visit
* Experienced severe hypoglycemia (Level 3 as defined in the ADA Standards of Medical Care in Diabetes (ADA 2022) within 3 months prior to the Screening Visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2023-10-19 (Actual); Primary Completion 2025-07-09 (Actual); Study Completion 2025-07-09 (Actual)

PRIMARY OUTCOMES:
Compare the effect of CT-868 versus placebo on change in HbA1c (%) from baseline | at Day 1 to Week 16

SECONDARY OUTCOMES:
Compare the effect of CT-868 versus placebo on change in HbA1c (%) from baseline | at Day 1 to Weeks 4, 8, and 12
To assess the percentage of participants achieving HbA1c of <7.0%. | at Week 16
To assess the percentage of participants achieving HbA1c of ≤6.5%. | at Week 16
To assess the percentage of participants achieving HbA1c of <5.7%. | at Week 16
Change in body weight (in kilograms) from baseline when comparing CT-868 to placebo. | at Day 1 to Week 16
Change in insulin doses from baseline when comparing CT-868 to placebo. | at Day 1 to Weeks 8 and 16

OTHER OUTCOMES:
Time In Range (TIR) as per Continuous Glucose Monitoring (CGM) metrics. | at Day 1 to Week 16
Time in hypoglycemia as per CGM metrics. | at Day 1 to Week 16
Time in hyperglycemia as per CGM metrics. | at Day 1 to Week 16

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Carmot Therapeutics, Inc., a member of the Roche Group
Locations (22):
- United States (22):
  - John Muir Physician Network Clinical Research Center, Concord, California
  - Headlands Research- AMCR, Escondido, California
  - University of Colorado - Barbara Davis Center for Diabetes, Aurora, Colorado
  - Denver Endocrinology Diabetes and Thyroid Center, Englewood, Colorado
  - Advent Health, Orlando, Florida
  - Orlando Health Science Clinic, LLC, Orlando, Florida
  - Innovative Research Institute, Port Charlotte, Florida
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - Rocky Mountain Clinical Research, LLC- Idaho Falls, Idaho, Idaho Falls, Idaho
  - Iowa Diabetes and Endocrinology Research Center, West Des Moines, Iowa
  - MedStar Health Research Institute - Washington Hospital Center, Hyattsville, Maryland
  - University of North Carolina Health Sciences at MAHEC, Asheville, North Carolina
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Lucas Research, Inc, Morehead City, North Carolina
  - Oregon Health and Science University, Portland, Oregon
  - Texas Diabetes and Endocrinology, P.A, Austin, Texas
  - Velocity Clinical Research - Dallas, Dallas, Texas
  - Research Institute of Dallas, Dallas, Texas
  - Diabetes & Glandular Disease Clinic, P.A., San Antonio, Texas
  - Consano Clinical Research, Shavano Park, Texas
  - Texas Valley Clinical Research, LLC, Weslaco, Texas
  - Rainier Clinical Research Center, Renton, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://carmot.us/